CLINICAL TRIAL: NCT02590198
Title: Diagnostic Performance Comparison Between Procalcitonin-based vs. ANAES-based Guidelines; Impact on Antibiotic Use in Newborns With Suspected Early-onset Neonatal Infection (EONI)
Brief Title: Diagnostic Performance Comparison Between Procalcitonin-based vs. ANAES-based Guidelines
Acronym: DIACORD
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: University Hospital, Tours (Other); University Hospital, Brest (Other); Rennes University Hospital (Other); Poitiers University Hospital (Other); University Hospital, Angers (Other Government); University Hospital, Bordeaux (Other); Centre Hospitalier de Bretagne Sud (Other); University Hospital, Paris (Other); Créteil Hospital (Other); Nantes Polyclinic (Unknown)
Responsible Party: Sponsor
Other Study IDs: RC15_0063
Record Dates: First submitted 2015-10-12; First posted 2015-10-28 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Early-onset Neonatal Infection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ANAES algorithm: Each center will start the study by applying the usual ANAES algorithm. The date of implementation of the new algorithm based on PCT will be determined randomly. Therefore, within each center, there will be an initial period in which the standard algorithm is applied and a second one during which the PCT-based algorithm is applied
  Interventions: Other: ANAES algorithm; Other: PCT algorithm
- PCT algorithm: Each center will start the study by applying the usual ANAES algorithm. The date of implementation of the new algorithm based on PCT will be determined randomly. Therefore, within each center, there will be an initial period in which the standard algorithm is applied and a second one during which the PCT-based algorithm is applied
  Interventions: Other: ANAES algorithm; Other: PCT algorithm

INTERVENTIONS:
Other: ANAES algorithm — care as recommended by ANAES, with ANAES algorithm
Other: PCT algorithm — care based on PCT algorithm

SUMMARY:
Neonatal bacterial infection remains a serious pathology in industrialized countries despite the use of prophylaxis measures for group B streptococcus (GBS) (peri-partum antibiotic in women with GBS colonization), which was implemented in the United States in 1996 and in France in 2001 and has led to a dramatic decrease in the incidence of neonatal bacterial infections. However, early onset neonatal infection (EONI), which is defined as an infection occurring during the first 6 days after birth (as opposed to late onset neonatal infections (LONI) occurring between days 7-89), is still one of the leading causes of neonatal morbidity and mortality. Physicians consider EONI a significant diagnostic and therapeutic emergency due to the potential for sudden onset and rapid evolution of sepsis in newborns with immature immune systems. Currently, in France, detection of EONI is based on national consensus guidelines published in 2002 (ANAES recommendations). There are broad indications to provide empirical antibiotic treatment pending diagnostic confirmation through different complementary exams. To ensure that every infected newborn is diagnosed, biological assessments are often repeated and result in the use of invasive and painful procedures, anemia and financial concerns. Moreover, in cases of abnormal biological results, many newborns are subjected to intravenous (IV) antibiotic treatments requiring hospitalization and separation from their mother. However recent studies have shown that antibiotics can have a potentially deleterious effect on the neonatal digestive microbiota and result in the appearance of antibiotic-resistant bacteria, with possible long-term consequences on the health of the child.

Procalcitonin (PCT) is a calcitonin prohormone secreted from the parenchymal tissues. This marker of inflammation has been shown to be a valuable diagnostic marker for bacterial infection in adults and in children. It also seems to be a reliable marker for neonatal bacterial infection, which would make it useful in the detection of EONI. Because physiological levels of PCT vary during the first days of life, possibly due to postnatal intestinal bacterial colonization, levels of this marker are difficult to interpret in the early neonatal period. However, in a study of 2151 newborns with suspected EONI, Nicolas Joram et al. found that PCT obtained from the umbilical blood cord, prior to newborn intestinal colonization, bypasses this postnatal physiological peak of PCT and effectively constitutes a discriminant marker to distinguish between infected and healthy infants using a cutoff value of 0.6 ng/ml.

Subsequent to this pilot study, several studies on PCT in umbilical blood cord confirmed its good diagnostic performance for EONI, particularly when included in a diagnostic algorithm. This marker could contribute to a better estimation of EONI risk in order to limit the use of unnecessary complementary exams and prescription of antibiotics and their associated short- and long-term side effects in healthy newborns.

Therefore, in this study, the investigators propose to test the diagnostic value of a PCT-based algorithm in newborns suspected of having EONI. The investigators hypothesize that this algorithm is as efficient as those currently used (ANAES), but will limit coinciding biological exams and exposure to antibiotics during the neonatal period.

ELIGIBILITY:
Inclusion Criteria:

* All children born at > 36 weeks gestation in one of the 15 participating maternity or neonatology units and suspected having EONI according to the ANAES recommendations (clinical suspicion of chorioamnionitis, intrapartum maternal fever > 38°C, infected twin, spontaneous premature delivery at < 37 gestational weeks, prolonged rupture of membrane for > 12 hours, maternal group B Streptococcus colonization without full prophylactic antibiotic treatment, or signs of fetal asphyxia) will be included in the study.
* Oral Consent (Non Opposition).

Exclusion Criteria:

* Newborns will be considered ineligible if:
* Parental non opposition is not obtained, if the parents do not speak French, present severe dementia and/or cannot be reached on day 6.
* Nosocomial neonatal infection, severe congenital malformation or obstetrically explained neonatal asphyxia are diagnosed.
* Secondary parental opposition.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children included in the DIACORD study will be born at > 36 weeks gestation in one of the 15 participating maternity or neonatology units and suspected of EOSI according to the ANAES recommendations (clinical suspicion of chorioamnionitis; intrapartum maternal fever > 38°C, infected twin, spontaneous premature delivery at < 37 gestational weeks, prolonged rupture of membrane for > 12 hours, maternal colonization with group B Streptococcus without full prophylactic antibiotic treatment, or signs of fetal asphyxia).
Sampling Method: Probability Sample
Enrollment: 9201 (Actual)
Dates: Start 2016-05-03 (Actual); Primary Completion 2017-01-22 (Actual); Study Completion 2017-01-22 (Actual)

PRIMARY OUTCOMES:
Primary outcome is a composite outcome including: death from any cause, intensive care unit admission for any reason, disease-specific complications, diagnosis of EONI after maternity discharge, need for antibiotics with hospital readmission | 6 days after birth
  The primary noninferiority endpoint is a composite of overall adverse outcomes induced by EONI occuring within 6 days following birth. It includes death, Neonatal Intensive care Unit (NICU) admission, or hospital readmission. The investigators chose this primary endpoint because the French definition of EONI diagnostic is subjective, specifically in case of possible EONI in case of gastric fluid positivity, and is finally rarely objectivated. Moreover, the new PCT-based algorithm do not require any gastric fluid analysis and modify the usual French definition of possible EONI, impossible to use in this context. Focusing on serious adverse event outcomes seems a very pragmatic and efficient methodologic strategy.

SECONDARY OUTCOMES:
death | Day 6 and Day 90
  components of the primary outcome (death/NICU/rehospitalisation + antibiotics) will be considered independently, as is advised for a composite outcome.
NICU admission | Day 6 and Day 90
  components of the primary outcome (death/NICU/rehospitalisation + antibiotics) will be considered independently, as is advised for a composite outcome.
rehospitalisation in connection with antibiotic treatment | Day 6 and Day 90
  components of the primary outcome (death/NICU/rehospitalisation + antibiotics) will be considered independently, as is advised for a composite outcome.
Inter-period frequency comparison of secondary adverse effect (SAE) and adverse effect (AE) related to antibiotics. | Day 6 and Day 90
Number of blood samples induced by the 2 algorithms | Day 6 and Day 90
  EONI diagnostic exams frequency for EONI induced by the 2 algorithms (number of blood samples)
Number of newborns investigated by the 2 algorithms | Day 6 and Day 90
  EONI diagnostic exams frequency for EONI induced by the 2 algorithms ( number of newborns investigated).
Inter-period cumulated hospital stay length (including maternity stay) | Day 90
clinical and biological description of EONI and LONI | 12 months
  Description of EONI and LONI bacteriological epidemiology (No recent data in France and Europe): frequency, typology...

CONTACTS AND LOCATIONS:
Overall Officials: GRAS-LEGUEN Christele, PU-PH, Principal Investigator — Nantes University Hospital
Locations (14):
- France (14):
  - Angers University Hospital, Angers
  - Bordeaux University Hospital, Bordeaux
  - Brest University Hospital, Brest
  - Créteil Intercommunal Center, Créteil
  - Lorient Hospital, Lorient
  - Private clinic - Polyclinique de l'Atlantique, Nantes
  - La Pitié Salpétrière Hospital (AP-HP), Paris
  - Robert Debré Hospital (AP-HP), Paris
  - Trousseau Hospital (AP-HP), Paris
  - Saint Joseph Hospital, Paris
  - Poissy-Saint germain Hospital, Poissy
  - Poitiers University Hospital, Poitiers
  - Rennes University Hospital, Rennes
  - Tours University Hospital, Tours